CLINICAL TRIAL: NCT02427269
Title: UNC Barrett's Esophagus and Esophageal Cancer Biorepository
Brief Title: University of North Carolina (UNC) Barrett's Esophagus and Esophageal Cancer Biorepository
Acronym: BEECAB
Status: Enrolling by invitation | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0444
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Barrett's Esophagus; Esophageal Cancer; Intramucosal Adenocarcinoma
Keywords: Barrett's Esophagus; Esophageal Cancer; Intramucosal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 1 10mL red tube and 1 8.5mL yellow tube for serum, plasma, and buffy collection
  * Up to 10 research-specific biopsies (tissue samples) obtained from the esophagus during the routine care EGD.
  * Pathology slides from routine care biopsies taken during the procedure as well as retrospective pathology slides from routine care biopsies taken prior to enrollment on the study.
  * Up to 4 cytology brushes during the procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Barrett's Esophagus (BE) Surveillance: Patients who have never received ablative therapy for Barrett's Esophagus and are receiving routine care surveillance upper endoscopy for their condition. Subjects will have esophageal biopsies, blood, and data collected for this study.
  Interventions: Other: Specimen Collection
- Barrett's Esophagus (BE) Pre-Ablation: Patients who are receiving routine care upper endoscopy with ablative therapy for their Barrett's Esophagus for the first time. Subjects will have esophageal biopsies, blood, and data collected for this study.
  Interventions: Other: Specimen Collection
- Barrett's Esophagus (BE) Post-Ablation: Patients with a history of Barrett's Esophagus who are status post ablation and are receiving routine care follow-up EGD for their condition. Subjects will have esophageal biopsies, blood, and data collected for this study.
  Interventions: Other: Specimen Collection
- Esophageal Cancer(ECA/IMC): Patients with esophageal cancer who are receiving routine care upper endoscopy for their condition. Subjects will have esophageal biopsies, blood, and data collected for this study.
  Interventions: Other: Specimen Collection
- Squamous Cell Carcinoma (SCC): Patients with squamous cell cancer of the esophagus who are receiving routine care upper endoscopy for their condition. Subjects will have esophageal biopsies, blood, and data collected for this study.
  Interventions: Other: Specimen Collection

INTERVENTIONS:
Other: Specimen Collection — * 1 10mL red tube and 1 8.5mL yellow tube for serum, plasma, and buffy collection
  * Up to 10 research-specific biopsies obtained from the esophagus during the routine care EGD.
  * Four biopsies will be taken from the midpoint of the current BE (or midpoint of previous BE if the patient has already received ablation for previous BE),
  * Two biopsies from normal squamous epithelium, and
  * One biopsy from each area of esophageal nodularity seen during the procedure
  * Pathology slides from routine care biopsies taken during the enrollment procedure, as well as retrospective pathology slides from routine care biopsies taken prior to enrollment on the study.
  * Up to 4 cytology brushes during the procedure.

SUMMARY:
Aim 1: To develop a prospective tissue and blood biorepository from patients with a history of Barrett's Esophagus (BE) or esophageal cancer (ECA) presenting to UNC hospitals for routine care upper endoscopy for their condition.

Aim 2: To collect clinical data from patients with a history of Barrett's Esophagus (BE) or esophageal cancer (ECA) that includes demographic data, endoscopic procedure data, and pathology data.

Aim 3: To integrate Aim 1 and 2 in a manner that will provide an efficient bi-directional flow of clinical information and specimens between laboratory and clinical scientists in order to foster innovative translational research.

Aim 4: To create a biorepository for future Institutional Review Board (IRB) approved studies that have tissue and/or blood specimen component.

DETAILED DESCRIPTION:
Patients will be identified during GI clinic visits or procedure visits with Dr. Nicholas Shaheen or his colleagues at UNC. Patients may also be identified by research personnel during review of the endoscopy schedule and medical records. If eligible, interested participants will be provided with a consent form during their clinic or procedure visit. Enrolled subjects will be assigned a unique identification (ID) number for data collection.

Patients will be recruited by Dr. Nicholas Shaheen and his colleagues or by other study personnel prior to their routine care endoscopy at UNC. An investigator, study coordinator, or other personnel trained in the protocol and referenced in the IRB application will obtain consent during the patient's visit in the GI clinic or prior to an upper endoscopy. Potential subjects will have an opportunity to carefully review the consent form, the details of the study will be reviewed verbally, and all questions will be answered to the satisfaction of the patient. Only English-speaking adults with the ability to consent will be eligible for enrollment in this study. After the subject signs the consent, a copy of the signed consent will be provided to the subject and the coordinator will collect demographic and historical information from the patient pertaining to illnesses, medication and other relevant information. The consent process will be documented in the subject's research file.

After obtaining informed consent, blood will be obtained and subjects will proceed with their routine care upper endoscopy. The endoscopist, as per routine practice, will note findings in the procedure report and photograph or record video to confirm and document key findings, as well as take biopsies as indicated for routine care. During the procedure up to 10 research biopsies will be collected as part of this study. Research biopsies will be collected in addition to routine care biopsies and will be obtained with a standardized biopsy protocol (below). The total number of research biopsies may vary based on presence/absence of nodularity but will not exceed 10 research-specific biopsies. This number of esophageal biopsies is within the standard of care for biopsying the esophagus.

Biopsies for clinical care are taken prior to any consideration of research biopsies. Research biopsies are taken only if the additional biopsies do not significantly increase the patient's risk or interfere with routine care procedures. The research biopsy protocol may be modified by the physician performing the procedure if necessary.

In addition to research blood and biopsies, up to 4 cytology brushings for research purposes may also be obtained during the procedure.

Specimens collected for this research study will include:

* 1 10mL red tube and 1 8.5mL yellow tube for serum, plasma, and buffy collection
* Up to 10 research-specific biopsies obtained from the esophagus during the routine care esophagogastroduodenoscopy (EGD).

  * Four biopsies will be taken from the midpoint of the current Barrett's Esophagus (BE) (or midpoint of previous Barrett's Esophagus (BE) if the patient has already received ablation for previous Barrett's Esophagus (BE)),
  * Two biopsies from normal squamous epithelium, and
  * One biopsy from each area of esophageal nodularity seen during the procedure
* Pathology slides from routine care biopsies taken during the procedure as well as retrospective pathology slides from routine care biopsies taken prior to enrollment on the study.
* Up to 4 cytology brushes during the procedure

Biopsies will be immediately frozen on liquid nitrogen then transferred to the -80 biorepository freezer for long term storage. Blood will be immediately processed and transferred to the -80 biorepository freezer for long-term storage.

The translational pathology lab (TPL) maintains formalin fixed paraffin embedded (FFPE) blocks from biopsies taken for routine care. Slides will be cut from these blocks for this study. Slide requests for this research study will not exhaust the archived tissue and will leave a substantial amount of the formalin fixed paraffin embedded (FFPE) block for potential future clinical use.

If subjects return for additional esophagogastroduodenoscopies (EGDs) as part of routine care, then all study procedures will be repeated as part of this registry as detailed below.

For subjects receiving routine care surveillance esophagogastroduodenoscopy (EGD) for current or previous Barrett's Esophagus (BE) or current or previous esophageal cancer (ECA): Specimens and data will be collected at each routine care surveillance EGD as part of this study.

For subjects receiving routine care treatment EGD for current BE/ECA: Specimens and data will be collected at the initial treatment EGD, but not during subsequent treatment EGDs. Once treatment is complete and BE or ECA is clear, this group will begin surveillance EGDs as part of routine care for their condition. Specimens and data will be collected during subsequent follow-up surveillance EGDs after treatment is complete.

Optional Additional Specimen Collection BEECAB participants who undergo ablative therapy will be followed to see whether they achieve CE-IM and those who achieve CE-IM will be followed to detect recurrent intestinal metaplasia and neoplasia (LGD, HGD or EAC) within Barrett's esophagus. Optional additional cytology brushings and biopsy samples will be collected for future investigations from participants undergoing any form of EET and with low grade dysplasia (LGD), high grade dysplasia (HGD), or intramucosal or T1a cancer and BE length > 1 cm. Those who had prior oncologic therapy with chemotherapy or radiation for esophageal cancer and have depth of cancer > T1a or metastatic disease will not be approached for additional samples.

Up to three research cytology brushings and 7 research forceps biopsy samples will be collected during their standard of care EGD for this optional specimen collection.

a) Patients with HGD, LGD, or ECA undergoing Endoscopic Therapy for the first time (initial EGD).

1. One cytology brushing from squamous tissue in the esophagus
2. Two cytology brushings from Barrett's Esophagus tissue
3. Up to five forceps biopsies from Barrett's Esophagus tissue
4. Up to two forceps biopsies from squamous tissue in the esophagus

b) Patients who have had prior ablation.

1. Up to two cytology brushings from neosquamous tissue in the esophagus post ablation
2. Up to two forceps biopsies from neosquamous tissue in the esophagus post ablation
3. Up to two forceps biopsies from squamous tissue in the esophagus
4. Up to two forceps biopsies from gastric fold

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and older.
* Able to read, comprehend, and complete the informed consent form.
* Presenting to UNC hospitals for routine care upper endoscopy for their condition.
* Meet one of the following:

  1. Current or previous diagnosis of Barrett's Esophagus (BE) with or without dysplasia OR
  2. Current or previous diagnosis of esophageal cancer (including esophageal adenocarcinoma, intramucosal carcinoma, and squamous cell carcinoma)
* Willing to undergo biopsy and blood collection for research purposes.

Exclusion Criteria:

* Unable to read or understand English.
* Current incarceration.
* Current use of blood thinners such as coumadin, warfarin, clopidogrel, heparin and/or low molecular weight heparin (requires discontinuation of medication 5 days prior to and 6 days after esophagogastroduodenoscopy [EGD] and/or ensuring blood thinners have been stopped within an appropriate time frame for that specific agent and in accordance with standard clinical practice).
* Known bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are receiving routine care upper endoscopy at UNC and meet the eligibility criteria detailed below.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-04-28 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Specimen Biorepository | 10 years
  To develop a prospective tissue and blood biorepository from patients with a history of Barrett's Esophagus (BE) or esophageal cancer (ECA) presenting to UNC hospitals for routine care upper endoscopy for their condition.
  To create a biorepository for future IRB approved studies that have a tissue and/or blood specimen component.
Data | 10 years
  To collect clinical data from patients with a history of Barrett's Esophagus (BE) or esophageal cancer (ECA) that includes demographic data, endoscopic procedure data, and pathology data.
Collaboration with other investigators | 10 years
  integrate Aim 1 and 2 in a manner that will provide an efficient bi-directional flow of clinical information and specimens between laboratory and clinical scientists in order to foster innovative translational research.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States